CLINICAL TRIAL: NCT01961986
Title: Rotator Cuff Sparing Total Arthroplasty - A Prospective, Randomized Clinical Trial
Brief Title: Rotator Cuff Sparing Total Arthroplasty
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 10-02125
Record Dates: First submitted 2013-10-08; First posted 2013-10-14 (Estimated); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Osteoarthritis; Inflammatory Arthritis
Keywords: Rotator Cuff; Rotator Cuff Sparing; Shoulder Replacement; Total Shoulder Replacement; Total Shoulder Arthroplasty; Arthritis
MeSH Terms: conditions — Osteoarthritis; Arthritis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TSR: traditional subscap release (Active Comparator): TSR - traditional subscapularis release approach
  Subscapularis tendon release technique TSR
  Interventions: Procedure: TSR - traditional subscapularis release
- TSR: rotator cuff sparing (Experimental): Rotator cuff sparing technique TSR
  Interventions: Procedure: TSR - rotator cuff sparing

INTERVENTIONS:
Procedure: TSR - traditional subscapularis release — Total Shoulder Replacement surgery performed using the traditional subscapularis release approach.
  Arms: TSR: traditional subscap release
Procedure: TSR - rotator cuff sparing — Total Shoulder Replacement surgery performed using the rotator cuff sparing approach.
  Arms: TSR: rotator cuff sparing

SUMMARY:
Design: Prospective, randomized clinical trial, of 120 patients requiring a total shoulder replacement (TSR).

Purpose: To collect and evaluate long-term clinical data on patients whose total shoulder replacement (TSR) is performed using the traditional surgical approach (called the subscapularis release approach) as compared to patients who have a TSR procedure done using a newer surgical approach (called the rotator cuff sparing approach).

DETAILED DESCRIPTION:
Design: Prospective, randomized clinical trial, of 120 patients requiring a total shoulder replacement (TSR).

Purpose: To collect and evaluate long-term clinical data on patients whose total shoulder replacement (TSR) is performed using the traditional surgical approach (called the subscapularis release approach) as compared to patients who have a TSR procedure done using a newer surgical approach (called the rotator cuff sparing approach).

For patients with arthritis, TSR can successfully improve pain and restore function. As a result, TSR has become the treatment of choice for patients with shoulder arthritis. Despite these generally good outcomes, however, there are concerns that rotator cuff function is suboptimal after surgery. One of the rotator cuff tendons is usually cut during the TSR procedure to insert the prosthesis and then repaired at the end of the surgery. If the tendon does not heal adequately, patients may experience persistent weakness, pain, and even failure of the replacement. Recently, a surgical technique called rotator cuff sparing TSR has been described where the procedure can be performed without ever cutting any of the rotator cuff tendons. As such, there should be minimized risk to the rotator cuff function after the surgery. Our study proposes to enroll two groups of patients with shoulder arthritis. The first group will be treated with the traditional TSR procedure. The second group will be treated with this new rotator cuff sparing surgical technique for TSR where the rotator cuff is never violated. After surgery, we will examine motion, strength, and functional use of the shoulder. In addition, we will specifically test the rotator cuff strength after the surgery. In this fashion, we plan to test the hypothesis that rotator cuff sparing TSR can improve the rotator cuff function while maintaining the excellent pain relief and motion that is normally observed after the traditional TSR procedure.

Enrollment: A total of approximately 120 subjects will be enrolled and treated at NYU Hospital for Joint Diseases. Subjects participating in the study will be randomly assigned to have their total shoulder replacement done using the traditional surgical approach (called the subscapularis release approach) or by the newer surgical approach (called the rotator cuff sparing approach). For each patient, a number will be created by a random number generator. Patients randomized to the even number (2) will receive a traditional TSA procedure that includes incision and repair of the subscapularis tendon during the procedure. Patients randomized to the odd number (1) will receive the rotator cuff sparing TSA. Regardless of the procedure, patients will remain "blind" to the type of procedure they received until completion of their 2 year follow up.

Follow-Up Requirements: Office Visits: Patients' participation will involve five (5) office visits (after surgery) over a period of two (2) years. At each visit, as part of the patients' regular care, they will have standard x-rays of their shoulder. All patients will complete self-administered questionnaires to assess the clinical outcome of the surgery and patients satisfaction. The patient administered outcome questionnaires will include the SF-12, and Patient Assessment Case Report Form.

ELIGIBILITY:
Inclusion Criteria:

* Patient is indicated for shoulder joint replacement
* Patient is at least 21 years of age
* Patient is expected to survive at least 2 years beyond surgery
* Patient is willing to participate by complying with pre-and post-operative visit requirements
* Patient is willing and able to review and sign a study informed consent form

Exclusion Criteria:

* Prior arthroplasty in the affected shoulder.
* Significant deformity of the proximal humerus that requires a custom made implant or where osteotomy of the shaft and / or the tuberosity has to be considered.
* Significant medial erosion of the glenoid such that lateral edge of the humeral head lies medial to the lateral rim of the acromion.
* Significant injury to the brachial plexus
* Inability or unwillingness to participate in the post operative evaluation for the entire 24 months period.
* Pregnant and lactating women will be excluded

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2010-07 (Actual); Primary Completion 2017-05-04 (Actual); Study Completion 2027-05-04 (Estimated)

PRIMARY OUTCOMES:
Functional Outcome | Preoperatively
  Patient subjective and objective data will be collected for all patients using the Short Form 12 (SF-12)and Patient Assessment forms. From these forms, both American Shoulder and Elbow Society (ASES) outcome score and the Constant score can be derived to assess functional outcome. Additional data will also be collected specific to the integrity and the function of the subscapularis tendon that include the results of the "belly press" and the "lift off" test. They will be graded as "unable", "maintain against gravity", "maintain against resistance", and "full strength."

CONTACTS AND LOCATIONS:
Overall Officials: Young W Kwon, MD, PhD, Principal Investigator — NYU Hospital for Joint Diseases
Locations (1):
- NYU Hospital for Joint Diseases, New York, New York, United States

REFERENCES:
- [Background] Deshmukh AV, Koris M, Zurakowski D, Thornhill TS. Total shoulder arthroplasty: long-term survivorship, functional outcome, and quality of life. J Shoulder Elbow Surg. 2005 Sep-Oct;14(5):471-9. doi: 10.1016/j.jse.2005.02.009. PMID 16194737
- [Background] Khan A, Bunker TD, Kitson JB. Clinical and radiological follow-up of the Aequalis third-generation cemented total shoulder replacement: a minimum ten-year study. J Bone Joint Surg Br. 2009 Dec;91(12):1594-600. doi: 10.1302/0301-620X.91B12.22139. PMID 19949123
- [Background] Lo IK, Litchfield RB, Griffin S, Faber K, Patterson SD, Kirkley A. Quality-of-life outcome following hemiarthroplasty or total shoulder arthroplasty in patients with osteoarthritis. A prospective, randomized trial. J Bone Joint Surg Am. 2005 Oct;87(10):2178-85. doi: 10.2106/JBJS.D.02198. PMID 16203880
- [Background] Norris TR, Iannotti JP. Functional outcome after shoulder arthroplasty for primary osteoarthritis: a multicenter study. J Shoulder Elbow Surg. 2002 Mar-Apr;11(2):130-5. doi: 10.1067/mse.2002.121146. PMID 11988723
- [Background] Armstrong A, Lashgari C, Teefey S, Menendez J, Yamaguchi K, Galatz LM. Ultrasound evaluation and clinical correlation of subscapularis repair after total shoulder arthroplasty. J Shoulder Elbow Surg. 2006 Sep-Oct;15(5):541-8. doi: 10.1016/j.jse.2005.09.013. Epub 2006 Jul 27. PMID 16979047
- [Background] Miller BS, Joseph TA, Noonan TJ, Horan MP, Hawkins RJ. Rupture of the subscapularis tendon after shoulder arthroplasty: diagnosis, treatment, and outcome. J Shoulder Elbow Surg. 2005 Sep-Oct;14(5):492-6. doi: 10.1016/j.jse.2005.02.013. PMID 16194740
- [Background] Miller SL, Hazrati Y, Klepps S, Chiang A, Flatow EL. Loss of subscapularis function after total shoulder replacement: A seldom recognized problem. J Shoulder Elbow Surg. 2003 Jan-Feb;12(1):29-34. doi: 10.1067/mse.2003.128195. PMID 12610483
- [Background] Gerber C, Yian EH, Pfirrmann CA, Zumstein MA, Werner CM. Subscapularis muscle function and structure after total shoulder replacement with lesser tuberosity osteotomy and repair. J Bone Joint Surg Am. 2005 Aug;87(8):1739-45. doi: 10.2106/JBJS.D.02788. PMID 16085613
- [Background] Qureshi S, Hsiao A, Klug RA, Lee E, Braman J, Flatow EL. Subscapularis function after total shoulder replacement: results with lesser tuberosity osteotomy. J Shoulder Elbow Surg. 2008 Jan-Feb;17(1):68-72. doi: 10.1016/j.jse.2007.04.018. Epub 2007 Nov 19. PMID 18024179
- [Background] Lafosse L, Schnaser E, Haag M, Gobezie R. Primary total shoulder arthroplasty performed entirely thru the rotator interval: technique and minimum two-year outcomes. J Shoulder Elbow Surg. 2009 Nov-Dec;18(6):864-73. doi: 10.1016/j.jse.2009.03.017. Epub 2009 Jun 21. PMID 19540778
- [Background] Gerber C, Hersche O, Farron A. Isolated rupture of the subscapularis tendon. J Bone Joint Surg Am. 1996 Jul;78(7):1015-23. doi: 10.2106/00004623-199607000-00005. PMID 8698718
- [Background] Gerber C, Krushell RJ. Isolated rupture of the tendon of the subscapularis muscle. Clinical features in 16 cases. J Bone Joint Surg Br. 1991 May;73(3):389-94. doi: 10.1302/0301-620X.73B3.1670434.
- [Background] Tokish JM, Decker MJ, Ellis HB, Torry MR, Hawkins RJ. The belly-press test for the physical examination of the subscapularis muscle: electromyographic validation and comparison to the lift-off test. J Shoulder Elbow Surg. 2003 Sep-Oct;12(5):427-30. doi: 10.1016/s1058-2746(03)00047-8. PMID 14564261